CLINICAL TRIAL: NCT05032391
Title: Multicenter, Prospective, Randomized, Double-blind Placebo-controlled Clinical Study of the Efficacy and Safety of the Vaccine for Prevention of Rotavirus Infection Pentavalent Live With the Participation of Healthy Children
Brief Title: Reactogenicity, Safety and Immunological Efficacy of the Live, Pentavalent Rotavirus Vaccine in Childhood Immunization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Limited Liability Company Pharm Aid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTV 003/18
Record Dates: First submitted 2021-08-09; First posted 2021-09-02 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Rotavirus Infection
Keywords: rotavirus vaccine
MeSH Terms: conditions — Rotavirus Infections | interventions — Freeze Drying

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized double-blind, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: The present study was a double-blind, placebo-controlled study, i.e., neither the investigator nor the parent / adoptive parent of the child knew which particular drug was administered to a particular study participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The pentavalent rotavirus vaccine (live attenuated oral, freeze-dried) (Experimental): Live attenuated bovine-human [UK] reassortant rotavirus vaccine manufactured by the Serum Institute of India, Limited (SIIL). The pentavalent vaccine contains rotavirus serotypes G1, G2, G3, G4, and G9 (≥5.6 log10 FFU/serotype/dose). The vaccine is lyophilized and supplied with 2.5 ml of citrate bicarbonate buffer added for reconstitution before oral administration.
  Interventions: Biological: The pentavalent rotavirus vaccine (live attenuated oral, freeze-dried)
- Diluent is a sterile solution (Citrate Bicarbonate Buffer) (Placebo Comparator): Same constituents as the active vaccine but without the viral antigens; manufactured by SIIL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: The pentavalent rotavirus vaccine (live attenuated oral, freeze-dried) — Three times orally in a volume of 2.5 ml (1 dose)
  Other Names: Rota-V-Aid™
  Arms: The pentavalent rotavirus vaccine (live attenuated oral, freeze-dried)
Drug: Placebo — Three times orally in a volume of 2.5 ml (1 dose)
  Other Names: Diluent is a sterile solution (Citrate Bicarbonate Buffer)
  Arms: Diluent is a sterile solution (Citrate Bicarbonate Buffer)

SUMMARY:
The first multicenter prospective, randomized, double-blind, placebo-controlled clinical trial of the pentavalent live vaccine for RVI prevention was conducted in Russia among healthy infants aged 2 months at the time of the first vaccination.

DETAILED DESCRIPTION:
The study is a double-blind placebo-controlled prospective randomized, of efficiency and safety of Vaccine to prevent a rotavirus infection pentavalent live with the participation of healthy children" is carried out in the Russian Federation according to the Protocol of clinical trial No. RTB 003/18, requirements of the national legal system and the international rules of conduct of clinical trials (ICH GCP). The study was randomized of 100 children corresponding to inclusion criteria and not having criteria of non-inclusion, which in the ratio 1:1 were randomized in one of two groups. Children from Group 1 received a vaccine to prevent a rotavirus infection pentavalent live, is triple orally with interval not less than four weeks of 2.5 ml (1 dose). Children from Group 2 received a placebo not less than four weeks of 2.5 ml (1 dose) are triple orally with an interval. Three children (2 persons from Groups 1 and 1 person of Group 2) who were ahead of schedule finished participation in the research were immunized once.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female children at the age of 2 months at the time of the first vaccination with PI / PS, vaccinated according to age by the schedule of the National Calendar of Preventive Vaccinations of the Russian Federation;
2. Baby should be ≥ 37 weeks gestational age and birth weight ≥ 2500 g;
3. Children who do not have contraindications for vaccination (by the Protocol, according to medical history and clinical examination);
4. An Informed Consent Form for participation in the research, voluntarily and personally signed by the parent / adoptive parent of the child, before any of the research procedures;
5. Ability, in the researcher's opinion, of the parents / adoptive parents of the child to comply with the requirements of the Protocol (attendance of all scheduled Visits, completion of the Child Observation Diary, etc.).

Exclusion Criteria:

1. Orphans (except for officially adopted children) and children without parental care;
2. Child's gestational age <37 weeks and birth weight <2500 g;
3. Participation in any other clinical study;
4. Received or planned vaccination with any other rotavirus vaccine before enrollment in this study;
5. A history of diarrhea or blood in the stool or a violation of bowel movements in the last 14 days;
6. A history of chronic diseases of the gastrointestinal tract, history of intussusception of the intestine and congenital malformations of the gastrointestinal tract, predisposing to it, surgery on the abdominal organs;
7. Known sensitivity or allergy to any of the PI and PS components;
8. Serious post-vaccination reactions/complications disorders/defects associated with any previous vaccinations;
9. Any significant systemic disease (from the lungs, liver, kidneys, skin, cardiovascular system, gastrointestinal tract, endocrine system, immune system, nervous system, and cancer or autoimmune disease) that would jeopardize children's health or result in non-compliance with the Protocol;
10. Congenital or genetic disorders/defects;
11. Clinically significant abnormalities in laboratory parameters that go beyond the limits of the normal range identified at the Screening and may have a negative impact on the safety of the child's participation in the study;
12. Household contact with immunocompromised people or with an immunocompromised pregnant woman;
13. In the researcher's opinion, the child is not eligible for inclusion in the study, or the researcher is convinced that the parent / adoptive parent will not follow the Protocol's procedures;
14. Continuous use (more than 14 days from birth until inclusion in the study) of immunosuppressants or immunomodulators;
15. Continuous use (more than 14 days from birth until inclusion in the study) of steroid drugs at a dose of more than 0.5 mg/kg/day in terms of prednisone. The use of topical or inhaled steroids is permitted;
16. A history of proven hepatitis B, diphtheria, tetanus, whooping cough, poliomyelitis, hemophilic or pneumococcal infection;
17. Confirmed or suspected immunodeficiency condition (based on medical history);
18. Hereditary or congenital immunodeficiency (according to family history );
19. Administration of immunoglobulins or blood components from birth until inclusion and their planned administration during the study.

Ages: 60 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Geometric mean concentration (GMC) of IgA antibodies | From 28 days post-Dose 3 to 1 year of age
  Increased number of specific antibodies IgA after threefold administration of HPV in the 1st group was statistically significantly different from the diversity of the increase in IgA level in the placebo group.
Seroconversion rate | From 28 days post-Dose 3 to 1 year of age
  Seroconversion rate (with two, three, and quadruple antibody increases) in the Group those grafted with the study drug ranged from 79.17% to 83.33%, with data values of effectiveness indicator of the studied Vaccine for prevention rotavirus infection statistically significantly exceeded levels seroconversion in children from the Placebo Group.
Seroconversion factor | From 28 days post-Dose 3 to 1 year of age
  The multiplicity of the increase in antibody HRT in the Vaccine Group was 39.05, in the Pla cebo Group -2,80. This indicator in the Vaccine Vaccinated Group is also statistically significant exceeded the seroconversion factor in the Placebo Group.
Occurrence of unsolicited adverse events | Within the 31 days (Day 0 - Day 30) after the vaccine dose
  The association with the study product had 44 adverse events (22 adverse events in study participants from Group 1 and 22 adverse events in study participants from Group 2). All adverse events that had a connection with taking the test product, were recorded within the first 7 days after immunization and were a manifestation of reactogenicity.
Occurrence of serious adverse events | Within the 31 days (Day 0 - Day 30) after the vaccine dose
  No history has been detected since severe post-vaccine reactions/complications related to the previous vaccination, allergic reactions to vaccine components, or any prior immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Irina V. Feldblium, PhD, Study Director — Perm State Medical University named after Academician E.A. Wagner; Olga A. Rychkova, Dr. Sci, Study Director — Tyumen State Medical University
Locations (2):
- Russia (2):
  - Perm State Medical University named after Academician E.A. Wagner, Perm
  - Tyumen State Medical University, Tyumen